CLINICAL TRIAL: NCT04751383
Title: Phase 1 Trial of Hu5F9-G4 (Magrolimab) Combined With Dinutuximab in Children and Young Adults With Relapsed and Refractory Neuroblastoma or Relapsed Osteosarcoma
Brief Title: Testing the Combination of Two Immunotherapy Drugs (Magrolimab and Dinutuximab) in Patients With Relapsed or Refractory Neuroblastoma or Relapsed Osteosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-00913; NCI-2021-00913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PED-CITN-03 (Other: Pediatric Early Phase Clinical Trial Network); PED-CITN-03 (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH); UM1CA228823 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-02-12 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: High Risk Neuroblastoma; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Refractory Neuroblastoma; Resectable Osteosarcoma
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma | interventions — Specimen Handling; Biopsy; dinutuximab; Magnetic Resonance Spectroscopy; magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (magrolimab, dinutuximab) (Experimental): Patients receive magrolimab IV and dinutuximab IV on study. Patients also undergo CT, MRI, and blood sample collection on study, as well as bone marrow aspiration and biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Dinutuximab; Procedure: Magnetic Resonance Imaging; Biological: Magrolimab
- Arm B (magrolimab, dinutuximab, surgery) (Experimental): Patients receive magrolimab IV and dinutuximab IV on study. Patients with pulmonary osteosarcoma may undergo surgical resection of tumor after cycle 1. After surgery, these patients continue receiving magrolimab and dinutuximab on study. Patients also undergo CT, MRI, and collection of blood samples on study, as well as bone marrow aspiration and biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Dinutuximab; Procedure: Magnetic Resonance Imaging; Biological: Magrolimab; Procedure: Resection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Magrolimab — Given IV
  Other Names: Hu5F9-G4; ONO 7913; ONO-7913; ONO7913
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: Arm B (magrolimab, dinutuximab, surgery)

SUMMARY:
This phase I trial is to find out the best dose, possible benefits and/or side effects of magrolimab in combination with dinutuximab in treating patients with neuroblastoma that has come back (relapsed) or does not respond to treatment (refractory) or relapsed osteosarcoma. Magrolimab and dinutuximab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread. The combination of magrolimab and dinutuximab may shrink or stabilize relapsed or refractory neuroblastoma or relapsed osteosarcoma. In addition, this trial may help researchers find out if it is safe to give magrolimab and dinutuximab after surgery to remove tumors from the lungs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of Hu5F9-G4 (magrolimab) in combination with dinutuximab in children and young adults with relapsed/refractory (R/R) neuroblastoma (NBL) or relapsed osteosarcoma.

II. Determine the recommended phase 2 dose (RP2D) of Hu5F9-G4 (magrolimab) given in combination with dinutuximab in children and young adults.

III. Determine the safety and feasibility of administering Hu5F9-G4 (magrolimab) in combination with dinutuximab to patients that undergo pulmonary resection of metastatic osteosarcoma within three weeks of surgery.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics (PK) of Hu5F9-G4 (magrolimab) in children and young adults.

II. Evaluate the event free survival (EFS) in two cohorts of patients who are treated at the recommended phase 2 dose (RP2D) (measurable relapsed osteosarcoma and patients with pulmonary relapse undergoing resection) and compare to historical controls.

III. Observe and record anti-tumor activity. IV. Evaluate the overall response rate (ORR) of patients in the NBL cohorts (measurable R/R NBL and evaluable R/R NBL) and osteosarcoma patients (measurable relapsed osteosarcoma) in the expansion cohorts treated at the RP2D.

EXPLORATORY OBJECTIVES:

I. To explore biomarkers of response and resistance including genomic (CD47 expression, Fc receptor [FcR] polymorphisms, SIRPa polymorphisms, and KiR phenotype) and immunologic (dinutuximab human anti-chimeric antibody [HACA], magrolimab anti-drug antibody [ADA], peripheral and bone marrow immune subsets, and circulating cytokines).

II. To explore biomarkers of response in the tumor microenvironment through multiplexed ion beam imaging (MIBI) on resected tissue or archival tissues including comparison of pre- and post- treatment tumor tissues from patients undergoing staged resection of pulmonary osteosarcoma.

OUTLINE: This is a dose de-escalation study of magrolimab with fixed-dose dinutuximab followed by a dose-expansion study. Patients are assigned to 1 of 2 arms.

ARM A: Patients receive magrolimab intravenously (IV) and dinutuximab IV on study. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and blood sample collection on study, as well as bone marrow aspiration and biopsy throughout the trial.

ARM B: Patients receive magrolimab IV and dinutuximab IV on study. Patients with pulmonary osteosarcoma may undergo surgical resection of tumor after cycle 1. After surgery, these patients continue receiving magrolimab and dinutuximab on study. Patients also undergo CT, MRI, and collection of blood samples on study, as well as bone marrow aspiration and biopsy throughout the trial.

After completion of study treatment, patients are followed up at months 2, 4, 6, 9 and 12 and then yearly until year 5, or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of histologically or cytologically confirmed NBL or osteosarcoma
* Patients must have:

  * Relapsed/refractory high-risk neuroblastoma (NBL) (defined as disease recurrence after completion of therapy, progressive disease on therapy, or refractory disease during induction therapy) or
  * Relapsed osteosarcoma (relapsed after frontline therapy and/or there must not be any potentially curative treatment options available at the time of enrollment)
* Cohort B1: Confirmed neuroblastoma: measurable NBL/ganglioneuroblastoma (defined as those lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with cross sectional imaging (CT scan or MRI), or >= 10 mm with calipers by clinical exam). Chest x-ray cannot be used to determine eligibility. Lesions must be iobenguane (MIBG) positive, positron emission tomography (PET) avid (if patient has a history MIBG negative disease) or biopsy proven NBL/ganglioneuroblastoma
* Cohort B2: Evaluable NBL (MIBG and/or bone marrow disease only)
* Cohort B3: Measurable osteosarcoma (defined as those lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm (>= 1 cm) with cross sectional imaging (CT scan, MRI, or calipers by clinical exam). Chest x-ray cannot be used to determine eligibility
* Cohort B4: Patients with relapsed resectable pulmonary osteosarcoma who are scheduled for a surgical resection
* Note: Subjects will not have measurable disease due to recently resected pulmonary metastases. Investigational therapy must begin within three weeks of resection. Staged resections are permissible; investigational therapy will be administered in between resections. Patients should receive one cycle of investigational therapy in between resections but can receive additional cycles to accommodate the most appropriate surgical schedule as determined by the treating physicians. Every effort will be made to have at least half of this cohort (five of ten patients) be those requiring a staged resection
* There is no limit to the number of prior treatment regimens. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to initiation of study treatment. Acute toxicity of any previous therapy must have resolved to grade 1 or less or stabilized, unless specified elsewhere

  * Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of initiation of study treatment (6 weeks if prior nitrosourea)
  * Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim
  * At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic non-myelosuppressive regimen
  * At least 4 weeks must have elapsed since prior therapy with 131I-MIBG
  * Monoclonal antibodies: At least 3 weeks must have elapsed since prior therapy that included a monoclonal antibody. Patients who have received prior therapy with GD2 antibodies, regardless of response to therapy, will be eligible
  * At least 7 days must have elapsed since the last pharmacologic dose of systemic corticosteroids
* Arm A: Age >= 2 or < 18 years of age
* Arm B: Age >= 2 or =< 35 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2; Subjects > 16 years of age: Karnofsky >= 50%; Subjects =< 16 years of age: Lansky scale >= 50%
* Absolute neutrophil count >= 1,000/mcL
* Hemoglobin >= 9.5 g/dL, transfusion support acceptable
* Platelets >= 100,000/mcL, independent of transfusions
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN) for age (sum of conjugated and unconjugated)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN
* Creatinine =< institutional ULN OR glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Female patients of childbearing potential must not be nursing or planning to be pregnant and must have a negative urine or serum pregnancy test within 30 days before enrollment and within 72 hours before the first administration of study treatment

  * Note: Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential
* The effects of Hu5F9-G4 (magrolimab) monoclonal antibody on the developing human fetus are unknown and dinutuximab is known to be teratogenic. For this reason, female patients of childbearing potential must be willing to use one highly effective method of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study and continue for 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * Male patients who are sexually active with a woman of childbearing potential (WOCBP) and who have not had vasectomies must be willing to use a barrier method of contraception (condom plus spermicidal gel) and refrain from sperm donation during the study and for 4 months after the last dose of study treatment. If the partner is pregnant, male patients must use barrier method contraception (condom) during the study and for 4 months after the last dose of study treatment to prevent fetal exposure to study treatment
* All patients and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will be obtained according to local institutional policy
* Cardiac ejection fraction >= 45% or shortening fraction >= 28%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO), multigated acquisition scan (MUGA) or cardiac MRI. No clinically significant electrocardiogram (ECG) findings that in the judgment of the treating investigator would present a contraindication for treatment

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-GD2 monoclonal antibody (dinutuximab) or Hu5F9-G4 (magrolimab) monoclonal antibody or other agents used in this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are receiving any other investigational agents
* Pregnant women are excluded from this study because Hu5F9-G4 (magrolimab) is a monoclonal antibody on the developing human fetus are unknown and dinutuximab may cause fetal harm. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Hu5F9-G4 (magrolimab) or dinutuximab, breastfeeding should be discontinued if the mother is treated with Hu5F9-G4 (magrolimab) or dinutuximab
* Patients who have received prior treatment with CD47 or SIRPalpha-targeting agents
* Patients with red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of RBCs transfused during the 4-week period prior to screening. RBC transfusions are permitted during the screening period and prior to enrollment
* Patients with known inherited or acquired bleeding disorders are not eligible
* Patients with prior hemolytic anemia or Evans syndrome in the last 3 months
* Patients with significant medical diseases that would worsen the risk-benefit ratio of participating in this study. This includes but is not limited to acute myocardial infarction within the last 6 months, unstable angina, significant acute or chronic infections, or severely immunocompromised state
* Patients on the following medications at the time of study treatment initiation:

  * Immunotherapy or immunosuppressive drugs (e.g. chemotherapy or systemic corticosteroids) EXCEPT for the following:

    * The only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product administration in order to avoid allergic transfusion reactions. The use of conventional doses of inhaled steroids for the treatment of asthma is permitted, as is the use of physiologic doses of steroids for patients with known adrenal insufficiency
  * Growth factors (granulocyte colony stimulating factor or granulocyte macrophage colony stimulating factor) EXCEPT for erythropoietin and darbepoietin alpha
  * Herbal remedies with immunostimulating properties (e.g., mistletoe extract) or known to potentially interfere with major organ function (e.g. hypericin)
* Patients administered a live vaccine within 28 days prior to initiation of study treatment
* Patients with active or previously treated central nervous system (CNS) metastasis

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robbie G Majzner, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (11):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two 'no treatment' patients were excluded from Arm A. There were zero patients assigned to Arm B/Expansion Cohort.
Groups:
- Arm A: Magrolimab 30 mg/kg: Dose Level 1: Participants were administered single agent Hu5F9-G4 (magrolimab) 30 mg/kg IV on day 1 of weeks 2 and 3 for a 21-day cycle safety lead-in cycle followed by Hu5F9-G4 (magrolimab) in combination with a fixed dose of dinutuximab in cycle 1 for up to a maximum of 12 cycles of combination therapy
- Arm A: Magrolimab 20 mg/kg: Dose Level -1: Participants were administered single agent Hu5F9-G4 (magrolimab) 20 mg/kg IV on day 1 of weeks 2 and 3 for a 21-day cycle safety lead-in cycle followed by Hu5F9-G4 (magrolimab) in combination with a fixed dose of dinutuximab in cycle 1 for up to a maximum of 12 cycles of combination therapy
- Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma: Expansion Cohort B1: Participants with confirmed neuroblastoma were administered a priming dose of Hu5F9-G4 (magrolimab) (1 mg/kg) on day 1 of week 1, RP2D followed by fixed dose of dinutuximab IV on days 2-5 of week 2, and RP2D on day 1 of week 3 and 4 for up to a maximum of 12 cycles of combination therapy
- Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma: Expansion Cohort B2: Participants with evaluable neuroblastoma were administered a priming dose of Hu5F9-G4 (magrolimab) (1 mg/kg) on day 1 of week 1, RP2D followed by fixed dose of dinutuximab IV on days 2-5 of week 2, and RP2D on day 1 of week 3 and 4 for up to a maximum of 12 cycles of combination therapy
- Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma: Expansion Cohort B3: Participants with measurable osteosarcoma were administered a priming dose of Hu5F9-G4 (magrolimab) (1 mg/kg) on day 1 of week 1, RP2D followed by fixed dose of dinutuximab IV on days 2-5 of week 2, and RP2D on day 1 of week 3 and 4 for up to a maximum of 12 cycles of combination therapy
- Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma: Expansion Cohort B4: Participants with resectable, pulmonary only relapsed osteosarcoma were administered a priming dose of Hu5F9-G4 (magrolimab) (1 mg/kg) on day 1 of week 1, RP2D followed by fixed dose of dinutuximab IV on days 2-5 of week 2, and RP2D on day 1 of week 3 and 4 for up to a maximum of 12 cycles of combination therapy
Period: Overall Study
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg | Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma | Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma | Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma | Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma
Started | 7 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two 'no treatment' patients were excluded from Arm A. There were zero patients assigned to Arm B/Expansion Cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg | Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma | Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma | Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma | Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma | Total
Number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 |  |  |  |  | 12
  Between 18 and 65 years | 0 | 0 |  |  |  |  | 0
  >=65 years | 0 | 0 |  |  |  |  | 0
Age, Continuous [Median (Full Range); unit: years] | 12.2 [6.6 to 16.8] | 11.9 [7.2 to 14.2] |  |  |  |  | 12.1 [6.6 to 16.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  |  |  |  | 1
  Male | 6 | 5 |  |  |  |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 |  |  |  |  | 2
  Not Hispanic or Latino | 5 | 2 |  |  |  |  | 7
  Unknown or Not Reported | 0 | 3 |  |  |  |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 |  |  |  |  | 1
  Asian | 0 | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  |  | 0
  Black or African American | 0 | 0 |  |  |  |  | 0
  White | 4 | 1 |  |  |  |  | 5
  More than one race | 1 | 1 |  |  |  |  | 2
  Unknown or Not Reported | 2 | 2 |  |  |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent (95% CI) of Participants With Grade 3 or Higher Adverse Events (Dose Finding Cohort)
Description: Percentage of evaluable patients experiencing grade 3 or higher adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 stratified by dose level.
Time Frame: Up to 30 days after last dose, maximum treatment duration 12 cycles (1 cycle = 21 days)
Population: 2 patients excluded as they did not receive treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg
Number analyzed (Participants) | 7 | 5
percentage of participants | 71.4 [29.0 to 96.3] | 100 [47.8 to 100]

2. Primary Outcome: Cycle 1 Dose Limiting Toxicities of Magrolimab
Description: Percent of DLT-evaluable subjects experiencing dose limiting toxicities during cycle 1 stratified by dose level.
Time Frame: During cycle 1 (21 days)
Population: There were 11 evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg
Number analyzed (Participants) | 6 | 5
percentage of participants | 33.3 [4.3 to 77.7] | 40 [5.3 to 85.3]

3. Primary Outcome: Percent (95% CI) of Participants With Grade 3 or Higher Adverse Events (Expansion Cohort)
Description: Percentage of evaluable patients experiencing grade 3 or higher AEs will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Within 3 weeks of surgery
Population: There were zero patients assigned to Arm B, therefore no data are available
Arm/Group | Arm B (Magrolimab, Dinutuximab, Surgery)
Number analyzed (Participants) | 0

4. Secondary Outcome: Serum Concentration Versus Time Curve of Hu5F9-G4
Description: Median (min, max) serum concentration versus time curve of Hu5F9-G4 (magrolimab) assessed at day 1, 8, and 15 of the safety lead in, day 1, 8, and 15 of cycle 1.
Time Frame: Assessed at day 1, 8, and 15 of the safety lead in, day 1, 8, and 15 of cycle 1
Population: All patients for whom PK were collected on a given timepoint are represented here. No samples collected from participants in the "Arm A: Magrolimab 20 mg/kg" Arm/Group during the Safety Lead-In day 8 and day 15
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg
Number analyzed (Participants) | 7 | 3
mcg/mL
  ARM A: Safety Lead-In day 1 (Week 1) | NA — concentrations too small to measure | NA — concentrations too small to measure
  ARM A: Safety Lead-In Day 8 (Week 2): number analyzed (Participants) | 3 | 0
  ARM A: Safety Lead-In Day 8 (Week 2) | NA — concentrations too small to measure |
  ARM A: Safety Lead-In Day 15 (Week 3): number analyzed (Participants) | 3 | 0
  ARM A: Safety Lead-In Day 15 (Week 3) | 214 [132 to 334] |
  ARM A:Cycle 1 Week 2 Day 1 | NA [upper limit 272] — concentrations too small to measure | NA — concentrations too small to measure
  ARM A:Cycle 1 Week 2 Day 8: number analyzed (Participants) | 6 | 2
  ARM A:Cycle 1 Week 2 Day 8 | 131 [13.3 to 312] | 52.2 [47.7 to 56.7]
  ARM A: Cycle 1 Week 3 Day 15: number analyzed (Participants) | 4 | 3
  ARM A: Cycle 1 Week 3 Day 15 | 357 [86.5 to 386] | 63 [upper limit 87.1] — concentrations too small to measure

5. Secondary Outcome: Percent (95% CI) of Responders Among Response-evaluable Participants
Description: Percent of response-evaluable patients with best response of partial response (PR) or complete response (CR) stratified by dose level.
Time Frame: Up to 3 years
Population: There were 11 evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg
Number analyzed (Participants) | 6 | 5
percentage of participants | 0 [0 to 45.9] | 0 [0 to 52.2]

6. Secondary Outcome: Event Free Survival (Expansion Cohort)
Description: The Kaplan-Meier method will be used to estimate 1-year event free survival (EFS) with 95% confidence interval as the time from study entry until relapse, secondary malignancy, or death.
Time Frame: Up to 1 year
Population: There were zero patients assigned to Arm B, therefore no data are available
Arm/Group | Arm B (Magrolimab, Dinutuximab, Surgery)
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Response Rate (Expansion Cohort)
Description: Percent of response-evaluable subjects with neuroblastoma with best response of complete response (CR) or partial response (PR) measured by Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: Up to 5 years post treatment
Population: There were zero patients assigned to Arm B, therefore no data are available
Arm/Group | Arm B (Magrolimab, Dinutuximab, Surgery)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose, maximum treatment duration 12 cycles (1 cycle = 21 days)
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Patients who didn't receive treatment are excluded from reporting of AEs.
Arm/Group | Arm A: Magrolimab 30 mg/kg | Arm A: Magrolimab 20 mg/kg | Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma | Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma | Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma | Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma
All-Cause Mortality (participants affected / at risk) | 5/7 | 2/5 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/7 | 5/5 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Magrolimab 30 mg/kg (N=7) | Arm A: Magrolimab 20 mg/kg (N=5) | Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma (N=0) | Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma (N=0) | Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma (N=0) | Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma (N=0)
Anemia (Blood and lymphatic system disorders) | 4 | 0 | NA | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 0 | 4 | NA | NA | NA | NA
Blood antidiuretic hormone abnormal (Investigations) | 0 | 1 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Dysphasia (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Edema cerebral (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Fatigue (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Fever (General disorders and administration site conditions) | 1 | 0 | NA | NA | NA | NA
Fever (General disorders and administration site conditions) | 0 | 2 | NA | NA | NA | NA
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | NA | NA | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 2 | 0 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 2 | NA | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 4 | 0 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 3 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | NA | NA | NA | NA
Pain (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 3 | 0 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 1 | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Serum sickness (Immune system disorders) | 1 | 0 | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA | NA | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
White blood cell decreased (Investigations) | 0 | 1 | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA | NA | NA
Disease progression (General disorders and administration site conditions) | 1 | 0 | NA | NA | NA | NA
Localized edema (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1 | NA | NA | NA | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Magrolimab 30 mg/kg (N=7) | Arm A: Magrolimab 20 mg/kg (N=5) | Arm B1: Magrolimab at the RP2D in Patients With Confirmed Neuroblastoma (N=0) | Arm B2: Magrolimab at the RP2D in Patients With Evaluable Neuroblastoma (N=0) | Arm B3: Magrolimab at the RP2D in Patients With Measurable Osteosarcoma (N=0) | Arm B4: Magrolimab at the RP2D in Patients With Resectable, Pulmonary Only Relapsed Osteosarcoma (N=0)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 1 | NA | NA | NA | NA
Alkaline phosphatase increased (Investigations) | 0 | 1 | NA | NA | NA | NA
Allergic reaction (Immune system disorders) | 1 | 0 | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 | 0 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 1 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA | NA
Bladder infection (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 2 | 0 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 3 | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | NA | NA | NA | NA
Blurred vision (Eye disorders) | 1 | 0 | NA | NA | NA | NA
Blurred vision (Eye disorders) | 0 | 1 | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
Capillary leak syndrome (Vascular disorders) | 2 | 0 | NA | NA | NA | NA
Capillary leak syndrome (Vascular disorders) | 0 | 1 | NA | NA | NA | NA
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | NA | NA | NA | NA
Cheilitis (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Chills (General disorders and administration site conditions) | 1 | 0 | NA | NA | NA | NA
Chills (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Creatinine increased (Investigations) | 2 | 0 | NA | NA | NA | NA
Creatinine increased (Investigations) | 0 | 2 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 3 | 0 | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 1 | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 1 | 0 | NA | NA | NA | NA
Edema face (General disorders and administration site conditions) | 0 | 2 | NA | NA | NA | NA
Eosinophilia (Blood and lymphatic system disorders) | 4 | 0 | NA | NA | NA | NA
Eosinophilia (Blood and lymphatic system disorders) | 0 | 3 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA | NA
Fatigue (General disorders and administration site conditions) | 4 | 0 | NA | NA | NA | NA
Fatigue (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Fever (General disorders and administration site conditions) | 6 | 0 | NA | NA | NA | NA
Fever (General disorders and administration site conditions) | 0 | 2 | NA | NA | NA | NA
Generalized edema (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Haptoglobin decreased (Investigations) | 1 | 0 | NA | NA | NA | NA
Headache (Nervous system disorders) | 4 | 0 | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 2 | NA | NA | NA | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 0 | NA | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0 | NA | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0 | NA | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3 | NA | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0 | NA | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | NA | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 3 | 0 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 2 | 0 | NA | NA | NA | NA
Lip pain (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Lipase increased (Investigations) | 1 | 0 | NA | NA | NA | NA
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 1 | 0 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 1 | NA | NA | NA | NA
Malaise (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | NA | NA | NA | NA
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 0 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 4 | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | NA | NA | NA | NA
Oral pain (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Pain (General disorders and administration site conditions) | 3 | 0 | NA | NA | NA | NA
Pain (General disorders and administration site conditions) | 0 | 1 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA | NA | NA | NA
Paresthesia (Nervous system disorders) | 0 | 2 | NA | NA | NA | NA
Penile pain (Reproductive system and breast disorders) | 1 | 0 | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Pharyngitis (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Photophobia (Eye disorders) | 0 | 1 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 3 | 0 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 2 | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 0 | 1 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 4 | 0 | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 3 | NA | NA | NA | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Thromboembolic event (Vascular disorders) | 1 | 0 | NA | NA | NA | NA
Thrush (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Upper respiratory infection (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 4 | 0 | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 2 | NA | NA | NA | NA
Ventricular tachycardia (Cardiac disorders) | 3 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Weight gain (Investigations) | 1 | 0 | NA | NA | NA | NA
Weight loss (Investigations) | 2 | 0 | NA | NA | NA | NA
Weight loss (Investigations) | 0 | 1 | NA | NA | NA | NA
White blood cell decreased (Investigations) | 4 | 0 | NA | NA | NA | NA
White blood cell decreased (Investigations) | 0 | 2 | NA | NA | NA | NA
Edema limbs (General disorders and administration site conditions) | 1 | 0 | NA | NA | NA | NA
Periorbital edema (Eye disorders) | 0 | 1 | NA | NA | NA | NA
Lung infection (Infections and infestations) | 0 | 1 | NA | NA | NA | NA
Dysesthesia (Nervous system disorders) | 0 | 1 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04751383/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04751383/ICF_002.pdf